CLINICAL TRIAL: NCT00833287
Title: Immunoregulatory Dysfunction in Trauma Patients: Role of Obesity
Acronym: ObesityRole
Status: Terminated | Type: Observational
Why Stopped: Enrollment process not efficient
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2008-0126
Record Dates: First submitted 2009-01-30; First posted 2009-02-02 (Estimated); Last update posted 2012-04-06 (Estimated); Status verified 2012-04

CONDITIONS: Trauma; Obesity
Keywords: immunoregulatory; dysfunction; obesity
MeSH Terms: conditions — Wounds and Injuries; Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No

SUMMARY:
Patient who have major traumatic injury are at risk to develop postoperative inflammatory complications such as pneumonia and lung trouble called adult respiratory distress syndrome (ARDS). This study will draw blood from trauma patients are several time points after their injury to see if we can predict who is at greatest risk for developing pneumonia or ARDS based upon the results of these immune lab tests. We are particularly interested to see if this will be useful in obese patients who have a greater risk of these post trauma complications

DETAILED DESCRIPTION:
The role of inflammation in disease is increasingly appreciated in clinical medicine. Too much or too long a course of inflammation can lead to serious and sometime fatal complications for patients who experience significant physical trauma, particularly those whose injuries are serious enough to warrant intensive care follow up. On the other hand, the sheer stress of the traumatic injury can leave patients deficient in their ability to mount a protective immune/inflammatory response leaving them susceptible to concomitant infection. Another component to the conundrum is that after the trauma (first hit), the surgeons are faced with the dilemma of complete surgical repair of the injury - the second hit (i.e. full orthopedic repairs) vs stabilization of the injury until the patient recovers from the shock of the first hit. The difficulty for the medical team is predicting who can safely tolerate a full second hit (total surgical restoration) vs who needs to be further stabilized before further intervention. In the obese individual, this conundrum is compounded by the known immune/inflammatory alterations characteristic of the obese state. How these patients in particular can be safely triaged for immediate vs delayed definitive therapy based upon specific immune/inflammatory parameters is the object of this initial pilot study.

Hypothesis

Obese individuals who experience severe traumatic injury will develop immunoregulatory dysfunction shortly after injury that is greater than nonobese individuals experiencing similar traumatic injury. Depending upon severity and duration of this immunoregulatory dysfunction, the post injury inflammatory responses will also be altered resulting in increased risk for pneumonia and/or adult respiratory distress syndrome, major morbidities associated with trauma.

Specific Aims

1. Determine immunoregulatory and inflammatory blood cytokine and endocrine stress hormone profiles in adult patients with significant traumatic injury correlated with subsequent development of pneumonia and/or adult respiratory distress syndrome.
2. Examine the role of obesity in the initial immunoregulatory dysfunction and subsequent short term clinical course of trauma patients.
3. Investigate whether demographic differences (age, gender, race) impact the risk for immunoregulatory and/or inflammatory dysfunction as well as risk for pneumonia and/or adult respiratory distress syndrome in obese s non obese trauma patients.

ELIGIBILITY:
Inclusion Criteria:

1. age 18 and older
2. traumatic injury of sufficient severity that ICU care is anticipated
3. Likely (by clinical criteria) to survive for at least 7 days after enrollment

Exclusion Criteria:

1. age less than 18 (not at risk for ARDS)
2. minor trauma not requiring ICU monitoring

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient with significant traumatic injury
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2008-11; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George V Russell, M.D., Principal Investigator — University of Mississippi Medical Center